CLINICAL TRIAL: NCT05089630
Title: A Phase 1/2, First-Time-in Human (FTiH), Randomized, Observer-blind, Placebo-controlled, Dose Escalation Study to Assess Safety, Reactogenicity and Immunogenicity of a Candidate Cytomegalovirus (CMV) Vaccine Comprising Recombinant Protein and Adjuvant When Administered Intramuscularly in Healthy Adults
Brief Title: A Study of Safety and Immune Response to Different Doses of a Cytomegalovirus Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 209976
Record Dates: First submitted 2021-10-11; First posted 2021-10-22 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Cytomegalovirus Infections
Keywords: Cytomegalovirus; First-Time-in Human; Safety; Reactogenicity; Immunogenicity; Healthy adults
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Pentamer(low)/gB(low)/Adjuvant Group (Experimental): Participants receive the candidate CMVsu vaccine consisting of a combination of low dose pentamer and low dose gB antigens, adjuvanted at 0, 2 and 6 months and are followed up until end of study (Day 546).
  Interventions: Biological: Pentamer (low)/gB(low)/Adjuvant vaccine
- Pentamer (med)/gB(low)/Adjuvant Group (Experimental): Participants receive the candidate CMVsu vaccine consisting of a combination of medium dose pentamer and low dose gB antigens, adjuvanted at 0, 2 and 6 months and are followed up until end of study (Day 546).
  Interventions: Biological: Pentamer (med)/gB(low)/Adjuvant vaccine
- Pentamer (med)/gB(med)/Adjuvant Group (Experimental): Participants receive the candidate CMVsu vaccine consisting of a combination of medium dose pentamer and medium dose gB antigens, adjuvanted at 0, 2 and 6 months and are followed up until end of study (Day 546).
  Interventions: Biological: Pentamer (med)/gB(med)/Adjuvant vaccine
- Pentamer (high)/gB(med)/Adjuvant Group (Experimental): Participants receive the candidate CMVsu vaccine consisting of a combination of high dose pentamer and medium dose gB antigens, adjuvanted at 0, 2 and 6 months and are followed up until end of study (Day 546).
  Interventions: Biological: Pentamer (high)/gB(med)/Adjuvant vaccine
- Placebo Group (Placebo Comparator): Participants receive placebo (saline) at 0,2 and 6 months and are followed up until end of study (Day 546).
  Interventions: Combination Product: Placebo (saline)

INTERVENTIONS:
Biological: Pentamer (low)/gB(low)/Adjuvant vaccine — Three doses of the candidate CMVsu vaccine consisting of a combination of low dose pentamer and low dose gB antigens, adjuvanted are administered intramuscularly in the deltoid region of the non-dominant arm in a 0, 2, 6-month schedule.
  Arms: Pentamer(low)/gB(low)/Adjuvant Group
Biological: Pentamer (med)/gB(low)/Adjuvant vaccine — Three doses of the candidate CMVsu vaccine consisting of a combination of medium dose pentamer and low dose gB antigens, adjuvanted are administered intramuscularly in the deltoid region of the non-dominant arm in a 0, 2, 6-month schedule.
  Arms: Pentamer (med)/gB(low)/Adjuvant Group
Biological: Pentamer (med)/gB(med)/Adjuvant vaccine — Three doses of the candidate CMVsu vaccine consisting of a combination of medium dose pentamer and medium dose gB antigens, adjuvanted are administered intramuscularly in the deltoid region of the non-dominant arm in a 0, 2, 6-month schedule.
  Arms: Pentamer (med)/gB(med)/Adjuvant Group
Biological: Pentamer (high)/gB(med)/Adjuvant vaccine — Three doses of the candidate CMVsu vaccine consisting of a combination of high dose pentamer and medium dose gB antigens, adjuvanted are administered intramuscularly in the deltoid region of the non-dominant arm in a 0, 2, 6-month schedule.
  Arms: Pentamer (high)/gB(med)/Adjuvant Group
Combination Product: Placebo (saline) — Three doses of placebo (saline) are administered intramuscularly in the deltoid region of the non-dominant arm in a 0, 2, 6-month schedule.
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to assess the safety, reactogenicity and immune response of the candidate CMV recombinant protein subunit (CMVsu) vaccine consisting of a combination of glycoproteins B (gB) and pentamer antigens adjuvanted, regardless of baseline CMV sero-status. This FTiH study will be conducted in healthy adults 18 to 50 years of age, in which the 4 dose levels of the vaccine will be administered in a step-wise dose escalation manner, based upon safety adjudication.

ELIGIBILITY:
Inclusion Criteria:

* Participants who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent obtained from the participant prior to performance of any study specific procedure.
* A healthy adult (woman or man), 18 to 50 years of age at the time of the first study intervention administration.
* Healthy participants as established by medical history and clinical examination before entering the study.
* Participants who are women of non-childbearing potential may be enrolled in the study.
* Participants who are women of child-bearing potential may be enrolled in the study, if the participant:

  * has practiced adequate contraception for 30 days prior to study intervention administration, and
  * has a negative pregnancy test on the day of study intervention administration and
  * has agreed to continue adequate contraception during the entire treatment period and for 3 months after completion of the study intervention administration series.
* Participants who agree to take appropriate infection control measures to prevent becoming infected with SARS-CoV2 during the study.
* Participants who initially fail screening due to COVID-19 infection may be re-screened and included in the study, within the screening window period.
* Participants with signs/symptoms suggestive of active COVID-19 (i.e., fever, cough, etc.) should be isolated for the time period recommended by CDC since the signs/symptoms started, and symptoms have resolved.
* Participants with known COVID-19 positive contacts should be quarantined for the time period since exposure recommended by CDC since the exposure and the participant remains symptom free or COVID test negative.
* Participants who are diagnosed with COVID-19 may receive their subsequent CMVsu vaccination dose provided they have no fever, and their condition is considered stable by the investigator (e.g., there may be mild lingering cough, but no shortness of breath or difficulty breathing) within the original schedule.
* Participants who initially fail screening due to other active infections may be re screened within the screening window period and included in the study, if they no longer have signs or symptoms of active infection in the judgment of the site investigator.
* If a participant has equivocal results on CMV serodiagnostic screening test, they are permitted to be re-screened if within the 60-day screening window. Flexibility in safety blood evaluations will be permitted within the Schedule of activities time intervals.

Exclusion Criteria:

Medical conditions

* Known documented medical history of or viral hepatitis B or C infection.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study intervention(s).
* Any confirmed or suspected immunosuppressive or immunodeficient condition.
* Family history of congenital or hereditary immunodeficiency.
* History of or current autoimmune disease.
* Lymphoproliferative disorder or malignancy within previous 5 years (excluding effectively treated non-melanotic skin cancer).
* Hypersensitivity to latex.
* Major congenital defects
* Acute or chronic clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality.
* Recurrent history or uncontrolled neurological disorders.
* Any hematological or biochemical abnormality.
* Any acute or chronic, clinically significant disease or pulmonary, cardiovascular, hepatic, or renal functional abnormalities.
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.
* Participants with symptoms suggestive of active COVID-19 infection are excluded.
* Participants with known COVID-19 positive contacts within the past 14 days should be excluded for at least 14 days since the exposure and the participant remains symptom free.
* Any other clinical condition that, might pose additional risk to the participant due to participation in the study.

Prior/Concomitant therapy

* Any history of or planned receipt of a CMV vaccine other than the study intervention at any time point.
* Use of other investigational/non-registered product during the period beginning 30 days before the first dose, or their planned use during the study period.
* Planned administration of any vaccine not foreseen by the study protocol 30 days before and 30 days after each study vaccination administration any licensed influenza vaccine administered > 15 days before/ after vaccination.
* In case of extraordinary emergency mass vaccination for an unforeseen public health threat the time period can be reduced if necessary, for that mass vaccination vaccine, which may be under emergency use authorization.

  * COVID-19 vaccines should be given at least 30 days before or after administration of a GSK study vaccine. This interval can be reduced to > 14 days, if emergency vaccination is recommended by public health authorities.
  * Candidate COVID-19 vaccines are not allowed.
* Chronic administration of immunosuppressants or other immune-modifying drugs within 3 months prior to the vaccine dose. Inhaled and topical steroids are allowed.
* Administration of long-acting immune-modifying drugs at any time during the study period.
* Administration of immunoglobulins and/or any blood products during the period starting 3 months before the administration of the first dose of study intervention(s) or planned administration during the study period.

Prior/Concurrent clinical study experience

• Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational intervention

Other exclusions

* Pregnant or lactating women. If a woman becomes pregnant/lactating during the study, she will be excluded from subsequent vaccine doses but will be followed for safety.
* Women planning to become pregnant or planning to discontinue contraceptive precautions before 3 months after last study vaccination.
* Participants with known high exposure risk for CMV transmission, to enable distinction of true vaccine effect from natural infection during the study.
* Planned move to a location that will prohibit participating in the trial until study end.
* Participants with current chronic alcohol consumption and/or drug abuse as defined by Diagnostic and Statistical Manual of Mental Disorders 5th edition.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 339 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
Number of participants reporting solicited administration site events | Within 7 days (the day of dose and 6 subsequent days) after each dose (vaccines administered on Day 1, Day 61 and Day 181)
  The solicited administration site events include pain, redness and swelling.
Number of participants reporting solicited systemic events | Within 7 days (the day of dose and 6 subsequent days) after each dose (vaccines administered on Day 1, Day 61 and Day 181)
  The solicited systemic events include fever, myalgia, fatigue, arthralgia and headache. The preferred location for measuring temperature is the oral cavity. Fever is defined as body temperature ≥38.0°C/100.4°F by any route.
Number of participants reporting unsolicited adverse events (AEs) within 7 days after each dose | Within 7 days (the day of dose and 6 subsequent days) after each dose (vaccines administered on Day 1, Day 61 and Day 181)
  An unsolicited AE is an AE that was not included in a list of solicited events using a Participant Diary. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms is reported as an unsolicited adverse event.
Number of participants reporting serious adverse events (SAEs) within 7 days after each dose | Within 7 days (the day of dose and 6 subsequent days) after each dose (vaccines administered on Day 1, Day 61 and Day 181)
  A SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant or is an abnormal pregnancy outcome.
Number of participants reporting unsolicited AEs up to 30 days after each dose | Up to 30 days after each dose (vaccines administered on Day 1, Day 61 and Day 181)
  An unsolicited AE is an AE that was not included in a list of solicited events using a Participant Diary. Unsolicited events must have been spontaneously communicated by a participant who has signed the informed consent. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms is reported as an unsolicited adverse event.
Number of participants reporting SAEs up to 30 days after each dose | Up to 30 days after each dose (vaccines administered on Day 1, Day 61 and Day 181)
  A SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant or is an abnormal pregnancy outcome.
Number of participants reporting medically attended AEs (MAEs) up to 30 days after each dose | Up to 30 days after each dose (vaccines administered on Day 1, Day 61 and Day 181)
  A MAE is an AE for which the participants received medical attention defined as hospitalization, an emergency room visit or a visit to or from medical personnel for any reason.
Number of participants reporting hematological and biochemical laboratory abnormalities on Day 1 | At Day 1
  The percentage of participants having hematology and biochemistry results below or above the laboratory normal ranges are tabulated by time point.
Number of participants reporting hematological and biochemical laboratory abnormalities on Day 8 | At Day 8
  The percentage of participants having hematology and biochemistry results below or above the laboratory normal ranges are tabulated by time point.
Number of participants reporting hematological and biochemical laboratory abnormalities on Day 61 | At Day 61
  The percentage of participants having hematology and biochemistry results below or above the laboratory normal ranges are tabulated by time point.
Number of participants reporting hematological and biochemical laboratory abnormalities on Day 68 | At Day 68
  The percentage of participants having hematology and biochemistry results below or above the laboratory normal ranges are tabulated by time point.
Number of participants reporting hematological and biochemical laboratory abnormalities on Day 181 | At Day 181
  The percentage of participants having hematology and biochemistry results below or above the laboratory normal ranges are tabulated by time point.
Number of participants reporting hematological and biochemical laboratory abnormalities on Day 188 | Day 188
  The percentage of participants having hematology and biochemistry results below or above the laboratory normal ranges are tabulated by time point.

SECONDARY OUTCOMES:
Number of participants reporting unsolicited AEs from Dose 1 to end of study (Month 18) | From Dose 1 (Day 1) to end of study (Month 18)
  An unsolicited AE is an AE that was not included in a list of solicited events using a Participant Diary. Unsolicited events must have been spontaneously communicated by a participant who has signed the informed consent. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms is reported as an unsolicited adverse event.
Number of participants reporting MAEs from Dose 1 to end of study (Month 18) | From Dose 1 (Day 1) to end of study (Month 18)
  A MAE is an AE for which the participants received medical attention defined as hospitalization, an emergency room visit or a visit to or from medical personnel for any reason.
Number of participants reporting SAEs from Dose 1 to end of study (Month 18) | From Dose 1 (Day 1) to end of study (Month 18)
  A SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant or is an abnormal pregnancy outcome.
Number of participants reporting potential immune-mediated disease (pIMDs) from Dose 1 to end of study (Month 18) | From Dose 1 (Day 1) to end of study (Month 18)
  PIMDs include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology.
Neutralizing antibodies (nAbs) titers against epithelial cell infection | On the day of each dose (Day 1, Day 61, Day 181), 30 days post each dose (Day 31, Day 91 and Day 211), 6- and 12-months post-Dose 3 (Day 361, Day 546)
  The humoral immune response is measured in terms of nAbs against epithelial cell infection and expressed as geometric mean titers (GMT). Serological assays for the determination of antibodies against CMV are performed by neutralization assay.
Anti-pentamer immunoglobulin G (IgG) and anti-gB IgG concentrations | On the day of each dose (Day 1, Day 61, Day 181), 30 days post each dose (Day 31, Day 91 and Day 211), 6- and 12-months post-Dose 3 (Day 361, Day 546)
  The vaccine-induced anti-gB and anti-pentamer humoral immune response is measured in terms of anti-pentamer IgG and anti-gB IgG geometric mean concentrations (GMCs) determined by enzyme linked immunosorbent assay (ELISA) and expressed in EU/ml.

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Hallandale, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Dearborn, Michigan
  - GSK Investigational Site, Springfield, Missouri
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, Secaucus, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Cedar Park, Texas
  - GSK Investigational Site, Galveston, Texas
  - GSK Investigational Site, Puyallup, Washington

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer tohttps://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

REFERENCES:
- [Derived] Sanchez-Martinez ZV, Alpuche-Lazcano SP, Stuible M, Durocher Y. CHO cells for virus-like particle and subunit vaccine manufacturing. Vaccine. 2024 Apr 11;42(10):2530-2542. doi: 10.1016/j.vaccine.2024.03.034. Epub 2024 Mar 19. PMID 38503664